CLINICAL TRIAL: NCT05682053
Title: Multiparametric MRI Imaging of Medullary Sponge Kidney
Brief Title: Multiparametric Magnetic Resonance Imaging (MRI) in Medullary Sponge Kidney
Acronym: MICARI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL22_0366; 2022-A01467-36 (Other: ANSM)
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Medullary Sponge Kidney
Keywords: medullary sponge kidney; kidney stone; multiparametric MRI; medullary function
MeSH Terms: conditions — Medullary Sponge Kidney; Kidney Calculi

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with medullary sponge kidney (Other): Patients with medullary sponge kidney attending medical consultation
  Interventions: Diagnostic Test: Multiparametic MRI
- Patients with glomerular filtration rate > 60 mL/min/1.73m2 without kidney stone (Other): Patients with glomerular filtration rate > 60 mL/min/1.73m2 without kidney stone attending a renal exploration.
  Interventions: Diagnostic Test: Multiparametic MRI

INTERVENTIONS:
Diagnostic Test: Multiparametic MRI — patients will have a Multiparametric MRI

SUMMARY:
Background :

Medullary sponge kidney disease is a congenital disorder caracterised by tubular ectasia and cystic dilatation of the collecting ducts in the pericalyceal region of the renal pyramids, which can lead to nephrolithiasis and frequently associated with impaired tubular function such as distal renal tubular acidosis.

The disease knowledge is limited, especially about origin, diagnosis, and physiopathology of the disease.

The disease is associated with impaired tubular function such as distal renal tubular acidosis, hypocitraturia, hypercalciuria, which suggest altered kidney medulla function.

Multiparametric MRI may provide further informations about the physiopathology and help in earlier diagnosis of the medullary sponge kidney.

Objective :

The aim of this study is to test the hypothesis that early kidney medulla function alteration in medullary sponge kidney can be detected and characterised with multiparametric MRI. We are expecting to see in medullary sponge kidney a decreased oxygenation content in BOLD MRI (Blood oxygenation level dependent magnetic resonance imaging), and decreased ADC (Apparent diffusion coefficient) value in the medulla.

Design :

A monocentric prospective case/control study will be conducted in adults with medullary sponge kidney. Controls are adults patients with glomerular filtration rate > 60 mL/min/1.73m2 without kidney stone attending a renal exploration.

After a screening visit, patients included will be evaluated on one day with lithiasis assessment and measurement of glomerular filtration (Urinary collection of the last 24 hours, Urine sample, Blood sample) and they will perform multiparametric magnetic resonance imaging of the kidneys.

ELIGIBILITY:
Inclusion Criteria:

* medullary sponge kidney attending medical consultation
* Patients with glomerular filtration rate > 60 mL/min/1.73m2 without kidney stone
* consent signed
* effective contraceptive method for women
* affiliated to social insurance scheme

Exclusion Criteria:

* kidney transplant
* polycystic kidney diseases
* Chronic kidney disease (GFR < 60 mL/min/1,73m² )
* MRI contraindications (claustrophobia, pacemaker, cardioverter defibrillators implantable, mechanical heart valve non MRI-compatible)
* Weight> 130 kg
* pregnancy
* legal protection measure (guardianship, curatorship)
* Deprived of liberty by a judicial or administrative decision
* subject participating in another research that may interfere with the research and including an exclusion period still in progress at inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Comparaison of R2* values measured by BOLD MRI beetween medullary sponge kidney patients and controls. | Day 0
  Comparaison of R2* values measured by BOLD MRI between medullary sponge kidney patients and controls.
  R2* is related to the level of tissue deoxyhemoglobin, which reflect tissue oxygenation.
  Increases in its outcome measure R2* (transverse relaxation rate expressed as per second) correspond to higher deoxyhaemoglobin concentrations and suggest lower oxygenation, whereas decreases in R2* indicate higher oxygenation.

SECONDARY OUTCOMES:
Comparaison of ADC value measured by diffusion-weighted MRI beetween medullary sponge kidney patients and controls. | Day 0
  Diffusion-weighted magnetic resonance imaging (DWI) is a non-invasive method sensitive to local water motion in the tissue, which is particularly sensitive to alterations in the renal interstitium, e.g. during renal fibrosis

OTHER OUTCOMES:
Comparaison of T1 Value measured by T1 mapping MRI between medullary sponge kidney patients and controls. | Day 0
  T1 mapping is a MRI sequence to estimate renal fibrosis
Comparaison of T2 Value measured by T2 mapping MRI between medullary sponge kidney patients and controls. | Day 0
  T2 mapping is a MRI sequence to estimate renal alteration
In medullary sponge kidney patients, evaluation of the association between kidney function and : - ADC value measured by diffusion-weighted MRI - T1 Value measured by T1 mapping MRI - T2 Value measured by T2 mapping MRI | Day 0
In medullary sponge kidney patients, evaluation of the association between 24 hours calciuria and : - ADC value measured by diffusion-weighted MRI - T1 Value measured by T1 mapping MRI - T2 Value measured by T2 mapping MRI | Day 0
  exploration if medulla modifications can lead to hypercalciuria
In medullary sponge kidney patients, evaluation of the association between 24 hours citraturia and : - ADC value measured by diffusion-weighted MRI - T1 Value measured by T1 mapping MRI - T2 Value measured by T2 mapping MRI | Day 0
  exploration if medulla modifications can lead to hypocitraturia
In medullary sponge kidney patients, evaluation of the association between urine pH and : - ADC value measured by diffusion-weighted MRI - T1 Value measured by T1 mapping MRI - T2 Value measured by T2 mapping MRI | Day 0
  exploration if medulla modifications is correlated to urine pH modifications
In medullary sponge kidney patients, evaluation of the association between maximum urinary osmolarity and : - ADC value measured by diffusion-weighted MRI - T1 Value measured by T1 mapping MRI -T2 Value measured by T2 mapping MRI | Day 0
  exploration if medulla modifications can lead to a decrease of renal concentration ability

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Result] Tournebize C, De Mul A, Abid N, Portefaix A, Pacaud S, Schleef M, Derain-Dubourg L, Rouviere O, Lemoine S. Medullary sponge kidney: in-depth phenotyping for a better understanding of functional and structural abnormalities. J Nephrol. 2025 Nov;38(8):2363-2373. doi: 10.1007/s40620-025-02413-3. Epub 2025 Sep 19. PMID 40973923